CLINICAL TRIAL: NCT03719482
Title: Assessment of the Biodistribution and Safety of [18F]MNI-1054 in Healthy Subjects
Brief Title: Assessment of the Biodistribution and Safety of [18F]MNI-1054
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-1054 Dosimetry
Record Dates: First submitted 2018-10-02; First posted 2018-10-25 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-1054 (Experimental): To measure blood metabolites of [18F]MNI-1054 in the healthy volunteers and to perform invasive as well as non-invasive modeling to assess its ability to measure LSD1 in the brain.
  Interventions: Drug: [18F]MNI-1054

INTERVENTIONS:
Drug: [18F]MNI-1054 — Healthy Volunteers recruited for the study will undergo a single [18F]MNI-1054 injection and PET scan.

SUMMARY:
The overall goal of this protocol is to evaluate the biodistribution of [18F]MNI-1054 as a LSD1 targeted radiopharmaceutical.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate the biodistribution of [18F]MNI-1054 as a LSD1 targeted radiopharmaceutical. The specific objectives are:

* To determine the radiation dosimetry of [18F]MNI-1054
* To assess the safety and tolerability of a single dose of [18F]MNI-1054

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and agree to participate by providing written informed consent.
* Are willing and able to comply with all study procedures and restrictions.
* Are males or females > 18 years of age and < 50 years of age.
* Are in good health as determined by the investigator based on clinical evaluations including past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening and prior to the first dose of study drug.
* Are a current nonsmoker who has not used tobacco- or nicotine-containing products (eg, nicotine patch) for at least 6 months prior to the first dose of study drug or first invasive procedure.
* Are a female subject of nonchildbearing potential, documented by medical records or physician's note to be either surgically sterile (by means of tubal ligation only) or post-menopausal for at least 1 year (i.e. 12 consecutive months with no menses without an alternative medical cause) or, if they are of childbearing potential, must commit to use two methods of contraception, one of which is a barrier method for the duration of the study.
* Are a male subject who is sterile or agrees to use an appropriate method of contraception, including a condom with or without spermicidal cream or jelly, from the first dose of study drug until 30 days after the last dose of study drug. No restrictions are required for a vasectomized male subject provided the subject is at least 1-year post bilateral vasectomy procedure prior to the first dose of study drug. A male subject whose vasectomy procedure was performed less than 1 year prior to the first dose of study drug must follow the same restrictions as a nonvasectomized man. Appropriate documentation of surgical procedure should be provided.
* Male subjects must not donate sperm for the study duration and for 30 days following the last dose of study drug.

Exclusion Criteria:

* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing. If needed (i.e. an incidental and limited need), acetaminophen is acceptable, but must be documented as a concomitant medication / significant non-drug therapy.
* Participation in any clinical investigation within four (4) weeks prior to initial dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines
* Has a known hypersensitivity to any component of the formulation of [18F]MNI-1054 or related compounds.
* Major surgery, or donation or loss of 400 mL or more of blood within four (4) weeks prior to initial dosing, or longer if required by local regulation.
* Have a history or presence of any significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders which, in the opinion of the investigator, are capable of altering the absorption, metabolism, or elimination of drugs or posing a health risk to participate in the study.
* The subject has a history of cancer (malignancy).
* Have clinically significant findings on laboratory evaluations.
* Have clinically significant findings on ECG evaluation.
* History of immunodeficiency diseases, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.
* History of drug or alcohol abuse within the 12 months prior to screening, or evidence of such abuse as indicated by the laboratory assays (i.e. positive drug or alcohol screen) conducted during the screening.
* The subject has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 oz], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
* The subject consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Positive pregnancy test result using serum beta-HCG, if female.
* Women who are lactating and breastfeeding.
* The subject is an employee of the sponsor or trial site or immediate family member (e.g., spouse, parent, child, sibling) of the sponsor or trial site.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Assessment of body organ distribution in Healthy Subjects | 2 months
  Whole body tomographic PET images will be obtained for 6 healthy volunteers, and reviewed visually for assessment of body organ distribution of radioactivity. Volumes of Interest (VOI) will be placed on the visually identified source organs, and subsequently used for all the study PET frames. Activity within these volumes of interest is expressed in units of total radioactivity (kBq).
  Radioactivity will be corrected for body attenuation, but not for decay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Madonia, PA-C, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://www.invicro.com